CLINICAL TRIAL: NCT05024565
Title: Prolonged Intravenous Infusion of β-lactam Antibiotics in Early Septic Patients
Acronym: PROBES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Wang Hao, associate professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Wang Hao
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Sepsis
Keywords: prolonged intravenous infusion; β-lactam Antibiotics; pharmacokinetics/pharmacodynamics (PK/PD)
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prolonged intravenous infusion of β-lactams Antibiotics (Experimental): Administer according to the PK/PD optimized regimen with the goal of increasing T>MIC. (1) Carbapenems: Calculate the daily dose according to the creatinine clearance rate and divide it into 3 times. Each time, the dose is injected intravenously at 1/2 dose for 15 minutes, and the remaining 1/2 dose is injected at a constant rate for 3 hours. (2) Cephalosporins: calculate the allowable daily dose according to the creatinine clearance rate, inject at a uniform rate within 24 hours. (3) β-lactams and β-lactamase inhibitor compound: the daily dose is calculated according to the creatinine clearance rate and injected at a uniform rate within 24 hours.
  Interventions: Behavioral: prolonged intravenous infusion of β-lactams Antibiotics
- short-term intravenous infusion of β-lactams Antibiotics (No Intervention): The daily allowable dose is calculated according to the creatinine clearance rate. The carbapenems, cephalosporins and β-lactamase inhibitor compound preparations are administered in accordance with the dosage and usage required by the instructions, and the injection is generally 30 minutes.

INTERVENTIONS:
Behavioral: prolonged intravenous infusion of β-lactams Antibiotics — (1) Carbapenems: Calculate the daily dose according to the creatinine clearance rate and divide it into 3 times. Each time, the dose is injected intravenously at 1/2 dose for 15 minutes, and the remaining 1/2 dose is injected at a constant rate for 3 hours. (2) Cephalosporins: calculate the allowable daily dose according to the creatinine clearance rate, inject at a uniform rate within 24 hours. (3) β-lactams and β-lactamase inhibitor compound: the daily dose is calculated according to the creatinine clearance rate and injected at a uniform rate within 24 hours.
  Arms: prolonged intravenous infusion of β-lactams Antibiotics

SUMMARY:
The prolonged β-lactam Antibiotics intravenous infusion strategy has emerged as the standard treatment for sepsis despite its unknown efficacy. The investigators will conduct a prospective, multi-center, cluster randomized controlled clinical trial. The investigators aimed to compare the clinical efficacy and prognosis of prolonged β-lactam antibiotics intravenous infusion versus short-term intravenous infusion in ICU patients with early sepsis. The investigators expect to recruit 40 branch centers and enroll at least 2600 patients with sepsis.

DETAILED DESCRIPTION:
Sepsis and septic shock can lead to high morbidity and mortality. The mortality of sepsis is related to inappropriate antibiotic treatment strategy. Due to the pathophysiological characteristics of patients with sepsis, the pharmacokinetics of antibiotics have changed, and antibiotic treatment strategies applied to general mild and severe infections may not be suitable for those patients. The relevant international guidelines recommend that antibiotic treatment for patients with sepsis should base on pharmacokinetic/pharmacodynamic principles, but this recommendation is based on low-level clinical evidence.

β-lactam antibiotics, including penicillins, cephalosporins, carbapenems and so on, are the most widely used antibacterial drugs in clinical practice. The best predictive parameter of those antibiotic bactericidal activity is the time during which the free drug concentration exceeds the target microbial MIC value (fT >MIC). According to Monte Carlo approach and clinical studies, as a PK/PD target value, an effective bactericidal effect can be achieved if fT>MIC reaches more than 40%; fT>MIC reaches more than 60%-70% can achieve the maximum bactericidal effect, which can be used in the treatment of severe cases. For severe infection and prevention of bacterial resistance, fT>MIC needs to reach 90%-100%.

The results of clinical studies have proved that improper or inadequate initial empiric antibiotic treatment is an independent risk factor that affects the therapeutic effectiveness and prognosis of severe infections. Important reasons for the lower-than-expected antibiotic treatment effect in severely ill patients include at least the following two factors: (1) Changes in the pathophysiological state of severely ill patients on drug metabolism, such as capillary leakage leading to increased drug distribution volume. As well as the high excretion and low obstruction hemodynamic characteristics of sepsis, increased renal blood flow leads to high excretion of water-soluble drugs, which often reduces the effective plasma concentration of the drug; (2) ICU infection of pathogenic bacteria has increased drug resistance and increased MIC. The above factors lead to the decrease of drug fT>MIC, which affects the efficacy of antibiotics. In recent years, the optimization of PK/PD-guided time-dependent antimicrobial treatment programs have confirmed that the administration method of prolonging the infusion time or continuous infusion can maintain a good steady-state blood drug concentration, prolong fT> MIC, and improve clinical curative effect, and can reduce the amount of antibiotics.

The main problems with PK/PD-guided antimicrobial therapy are: (1) Lack of convincing large sample clinical research results; (2) It has not been confirmed which subgroup (such as the sepsis severity, drug-resistant patterns of pathogens, immunocompetence) can be benefited from this strategy; (3) It is not clear whether the method of prolonged infusion can be applied in all kinds of β-lactam antibiotics .

This study adopts multi-center, openness, cluster randomization method to group, and eliminates the bias caused by factors such as the treatment environment in a single ward through the multi-center study; through Uniform training realizes the standardization of drug delivery methods to eliminate researchers' human bias in treatment operations and observations. At the same time, the regional randomization method sets the drug delivery method for a certain research center in a certain research phase to be determined, which eliminates the operational error and observation bias when the researcher needs to face multiple drug delivery programs at the same time. It can greatly reduce research costs and human bias, and more reliably obtain the impact of PK/PD-guided antibiotic treatment on the prognosis of patients and the impact of bacterial resistance in the entire ward.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in ICU who need to be treated with β-lactam antibiotics for clinical diagnosis of infection;
2. Meet the diagnostic criteria of sepsis 3.0 in the previous 24h;
3. At assessment of eligibility, treating doctor expects patient to need treatment in ICU beyond the next calendar day.

Exclusion Criteria:

1. The infection is diagnosed clinically, but the acquired pathogens are not sensitive to the study drug;
2. Has a history of allergies to study drugs;
3. Those who have a serious condition and the expected survival time is less than 72 hours.
4. Receipt of potential study medication for > 24 hours before randomization.
5. Pregnancy
6. Death is deemed imminent and inevitable.
7. Receiving palliative or supportive treatment only at the time of assessment for eligibility.
8. Treating doctor not committed to provision of advanced life-support, including any of mechanical ventilation, dialysis and vasopressor administration for at least the next 48 hours.
9. Consent not gained for study participation and entry under a waiver-of-consent not approved by the jurisdictional human research ethics committee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality in ICU | Change of mortality between two arms at 90-day from the day antibiotic therapy begin.
  Prolonged β-lactamase Antibiotics Infusion lower the All-cause mortality in ICU compared with normal group
28-day all-cause mortality | Change of mortality between two arms at 28-day from the day antibiotic therapy begin.
  Prolonged β-lactamase Antibiotics Infusion lower 28-day all-cause mortality the compared with normal group

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and ICF will be shared with other researchers when start this trial.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and ICF will be shared with other researchers when start this trial for five years.
Access Criteria: Ever researchers can access our study protocol and ICF from the web of clinical trials.gov.

DOCUMENTS (2):
  • Study Protocol (2021-08-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT05024565/Prot_000.pdf
  • Informed Consent Form (2021-08-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT05024565/ICF_001.pdf